CLINICAL TRIAL: NCT04185012
Title: NAsal Polyps: Inflammatory & Molecular Phenotyping of Responders to Benralizumab
Acronym: NAPPREB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Humanitas Clinical and Research Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NAPPREB
Record Dates: First submitted 2019-11-29; First posted 2019-12-04 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Nasal Polyps
Keywords: Benralizumab; Biomarkers; Eosinophils
MeSH Terms: conditions — Nasal Polyps | interventions — benralizumab

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled clinical trial. Patients will be divided in two arms with 1:1 randomization to Treatment or Placebo.
Who Masked: Investigator
Masking Description: Randomization will occur by assigning a unique sequential study code to a balanced number of randomly assorted treatment vials.
  An online open source randomization software will be used to assign treatment groups, and this will be done by an external person from those who will follow and treat the patients.
  Patients randomization will be blinded to the patients themselves and to all the personnel that will have contact with them during the trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Benralizumab (Experimental): Benralizumab 30 mg administered subcutaneously every 4 weeks for the first 3 doses and then every 8 weeks, for a treatment-period of 16 weeks
  Interventions: Biological: Benralizumab
- Placebo (Placebo Comparator): Placebo administered subcutaneously every 4 weeks for the first 3 doses and then every 8 weeks, for a treatment-period of 16 weeks
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Benralizumab — Benralizumab 30 mg administered subcutaneously Q4W for the first 3 doses and then Q8W, for a 16 weeks treatment-period
  Arms: Benralizumab
Biological: Placebo — Placebo administered subcutaneously Q4W for the first 3 doses and then Q8W, for a 16 weeks treatment-period
  Arms: Placebo

SUMMARY:
Background and rationale:

Phase III-b study.

Population and patient selection criteria: Adult patients with Chronic Rhinosinusitis with Nasal Polyps (allergic and non-allergic) requiring at least 1000 mg oral prednisone over the previous twelve months to control symptoms of rhinosinusitis, and with:

* Nasal polyps score (Meltzer et al.) ≥ 5
* Symptoms VAS scores (for nasal obstruction, hyposmia, post-nasal drip, sneezing, rhinorrea; 0-10 for each symptom) > 24 Sample size: 20 subjects.

Study design and study duration:

This is a pilot, prospective, double-blind placebo-controlled (DBPC) phase III-b trial with Benralizumab 30 mg administered subcutaneously every 4 weeks for the first 3 doses and then every 8 weeks, for a treatment-period of 16 weeks (followed up at 32 and 52 weeks) in patients with chronic rhinosinusinusitis with nasal polyps (CRSwNP).

Description of study treatment/product/intervention: Benralizumab, 30 mg subcutaneously every 4 week for the first 3 doses, and then every 8 weeks.

Objectives:

* Primary objective: To assess the clinical efficacy of Benralizumab on CRSwNP at week 24 (vs baseline) after the beginning of treatment, and to correlate the presence of baseline biomarkers with nasal polyp (NP) score improvement, in order to identify any possible predictive biomarker of response to Benralizumab.
* Secondary objective: In the follow up phase we will monitor all the biomarkers at 32 and 52 weeks , this monitoring will ascertain if any of those will predict relapse of nasal polyps and consequently when Benralizumab treatment has to be reinstalled.
* Safety objective: To evaluate the safety and tolerability of Benralizumab in patients with CRSwNP

Statistical methods, data analysis: Descriptive analysis of all collected variables at all time-points will be performed. Patients will be classified into "responders" and "non responders", for primary endopoint variable. Continuous variables will be evaluated with the normality test of Kolmogorov-Smirnov and compared with ANOVA or the Mann-Whitney test, depending on the normality of distribution. Categorical variables will be compared using Fisher's exact test.

Ethical considerations: The study will be performed in accordance with ethical principles that have their origin in the Declaration of Helsinki and are consistent with ICH/Good Clinical Practice, applicable regulatory requirements and the Sponsor policy on Bioethics and Human Biological Samples.

ELIGIBILITY:
Inclusion Criteria:

Adult patients with Chronic Rhinosinusitis with Nasal Polyps (allergic and non-allergic) requiring at least 1000 mg oral prednisone over the previous twelve months to control symptoms of rhinosinusitis, and with:

* Nasal polyps score (Meltzer et al.) > 5
* Symptoms VAS scores (for nasal obstruction, hyposmia, post-nasal drip, sneezing, rhinorrea; 0-10 for each symptom) > 24
* Provision of informed consent prior to any study specific procedure

Exclusion Criteria:

* Patients < 18 years age
* Pregnant women
* Biologic therapy in the past 6 months (or at least a period corresponding to 5 half-life of used drugs) (eg: omalizumab, mepolizumab, reslizumab, dupilumab)
* Previous treatment with Benralizumab
* Known hypersensitivity to benralizumab or any of its excipients
* Immunosuppression other than oral steroids in the past 3 months
* Allergen immunotherapy in the past 6 months
* Serious life threatening cardiopulmonary disorders
* Systemic immunologic disorder in the last 12 months
* Positive history for malignant tumors ever in patient's life
* Patients with conditions or concomitant diseases making them non evaluable at visit 1 or for the primary efficacy endpoint:

  1. Ongoing rhinitis medicamentosa
  2. Nasal septal deviation occluding at least one nostril
  3. Acute sinusitis, nasal infection, upper respiratory infections
  4. Radiologic suspicion or confirmed invasive or expansive fungal rhinosinusitis
  5. Eosinophilic Granulomatosis with Polyangiitis (previously named Churg-Strauss Syndrome)
  6. Granulomatosis with Polyangiitis (previously named Wegener's granulomatosis)
  7. Young's Syndrome
  8. Kartagener's Syndrome
  9. all ciliary dyskinesia
  10. Cystic Fibrosis
* Systemic corticosteroid treatment for other chronic conditions (i.e.: autoimmune disorders, tumors,….)
* Evidence of active systemic immunedepression (i.e..: primary or secondary immunodeficiency)
* Patients with severe asthma, defined according to ERS/ATS definition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Significant reduction of the Nasal polyps Score (range: 0-8; higher values mean larger nasal polyps size) | at week 24 (vs baseline)
  score reduction of 1.5

SECONDARY OUTCOMES:
Reduction in Lund-MacKay Score (range: 0-24; higher values mean larger nasal polyps extension) | at week 24 (vs baseline)
  >50% of baseline
Improvement of Sino-Nasal Outcome Test (SNOT-22; range: 0-110; higher values mean poorer disease-related quality of life) | at week 24 (vs baseline)
  >40% of baseline
Improvement of smell Visual Analogue Scale (VAS; range: 0-10; higher values mean worse smell) | at week 24 (vs baseline)
  >50% of baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Clinical and Research Hospital, Rozzano, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chong LY, Piromchai P, Sharp S, Snidvongs K, Webster KE, Philpott C, Hopkins C, Burton MJ. Biologics for chronic rhinosinusitis. Cochrane Database Syst Rev. 2021 Mar 12;3(3):CD013513. doi: 10.1002/14651858.CD013513.pub3. PMID 33710614